CLINICAL TRIAL: NCT02307448
Title: Effectiveness of Autologous Platelet Rich Plasma in the Treatment of Chronic Non-Healing Wounds
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of patient enrollment and lack of reimbursement
Sponsor: ACR Biologics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10312014
Record Dates: First submitted 2014-12-02; First posted 2014-12-04 (Estimated); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Foot Ulcer Chronic; Skin Ulcer Venous Stasis Chronic; Pressure Ulcer
MeSH Terms: conditions — Pressure Ulcer | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PRP Group (Active Comparator): Patients will receive weekly PRP treatments
  Interventions: Procedure: Platelet Rich Plasma
- Standard of Care (Placebo Comparator): Patients will receive weekly standard of care.
  Interventions: Procedure: Standard of Care

INTERVENTIONS:
Procedure: Platelet Rich Plasma — Patients will receive weekly PRP treatments with standard of care.
  Other Names: PRP
  Arms: PRP Group
Procedure: Standard of Care — Patients will receive weekly standard of care.
  Arms: Standard of Care

SUMMARY:
This investigation plans to initiate the healing of chronic wounds by providing a concentrated platelet and growth factor therapy directly to the wound site by topical delivery. This therapy will be derived from autologous platelet rich plasma (PRP), an emerging surgical and wound care treatment. This investigation aims to demonstrate that patients with chronic, non-healing wounds treated with autologous PRP and standard medical care have a reduction in wound volume and improved healing rate that results in patient-centered clinically significant health outcomes as compared to patients treated with standard medical care only.

DETAILED DESCRIPTION:
This is a multicenter randomized controlled trial, with a single-blind parallel design. 1,500 subjects are planned to enroll in the study. Each subject will be assigned to the treatments in random order. The stratified permuted block randomization method will be applied to the patient assignment. In addition to three study populations, i.e., DFU, VU and PU, and study centers, stratification will be based on one overall variable, (1) nutritional status (Low: Prealbumin <12mg/d vs. moderate: Prealbumin >= 12 mg/d) and one variable for each wound type. Diabetic food ulcer will be based on offloading (2a) (Specialty shoes vs. Total contact cast), pressure ulcer will be based on offloading (2b) (mattress vs. cushion), and venous leg ulcer will be based on compression (2c)(Low: <10 mmHG vs. High: >=30mmHG). Randomization will proceed within strata according to a permuted block scheme with a block size, or balancing interval, varying randomly between 2, 4 or 6. The primary endpoint will be evaluated by a blinded physician to avoid the bias.

Total duration of each patient in the study is expected to be 20 weeks.

ELIGIBILITY:
6.2 Inclusion Criteria

* Male or female ≥ 18 years of age.
* Wound must be diagnosed as Diabetic Foot Ulcers (DFU), Venous Ulcers (VU), or Pressure Ulcers (PU) with duration greater than 30 days at first visit/patient screening.
* If more than one non-healing wound is present, the largest wound will be selected and must be at least 2cm in size.
* Wound must be classified as Wagner 1 - 3 on the Wagner classification system. Wagner's Classification System Grade 1 Superficial ulcer without subcutaneous tissue involvement Grade 2 Penetration through the subcutaneous tissue (bone, tendon, ligament or joint capsule) Grade 3 Osteitis, abscess or osteomyelitis Grade 4 Gangrene of the forefoot Grade 5 Gangrene of the entire foot
* There must be at least 2 cm between the index wound and other wounds; if all wounds are closer than 2 cm, the patient should not be enrolled (screen failure).
* Wound must be clinically non-infected (A swab or deep tissue culture shall be performed at the discretion of the provider).
* If a female of childbearing potential, the patient must have a negative serum pregnancy test at screening.
* Patient has the capacity to understand and consent to be in the study. Written informed consent must be obtained from either the patient or the patient's legally acceptable representative prior to screening activities.
* Platelet count ≥ 75,000 (according to CBC)
* Hemoglobin (Hgb) level > 9 g/dL (according to CBC)
* Hematocrit (HCT or Ht) level > 27% (according to CBC)
* Ankle-Brachial Index (ABI) Test > 0.7

6.3 Exclusion Criteria

* Male or female <18 years of age
* Patients with known sensitivity to components of the PRP kit (calcium chloride, thrombin, collagen, acid citrate dextrose solution A (ACDA).
* Wound is not a Diabetic Foot Ulcers (DFU), Venous Ulcer (VU), or Pressure Ulcer (PU) at duration of greater than 30 days at first visit/patient screening.
* Wounds smaller than 2cm will be excluded. Exclusion criteria do not include maximum wound size or age.
* Wound that is classified as Wagner 4 - 5 on the Wagner classification system. Wagner's Classification System Grade 1 Superficial ulcer without subcutaneous tissue involvement Grade 2 Penetration through the subcutaneous tissue (bone, tendon, ligament or joint capsule) Grade 3 Osteitis, abscess or osteomyelitis Grade 4 Gangrene of the forefoot Grade 5 Gangrene of the entire foot
* There is less than 2 cm between the index wound and other wounds; if all wounds are closer than 2 cm, the patient should not be enrolled (screen failure).
* Wound is clinically infected. (A swab or deep tissue culture shall be performed at the discretion of the provider).
* Presence of non-treated osteomyelitis.
* If female, patient is pregnant, nursing or plans to become pregnant during the duration of the trial.
* Patients who are cognitively impaired and do not have a healthcare proxy.
* Platelet count < 75,000 (according to CBC)
* Hemoglobin (Hgb) level ≤ 9 g/dL (according to CBC)
* Hematocrit (HCT or Ht) level ≤ 27% (according to CBC)
* Ankle-Brachial Index (ABI) Test ≤ 0.7
* Patient has lymphedema.
* Received electrostimulation, hyperbaric treatments, systemic corticosteroids, growth factors or any cell or tissue derived products for any wounds 30 days prior to entry into the study. (Except for patients receiving inhaled corticosteroid treatments for COPD)
* Received radiation therapy or chemotherapy within previous 3 months.
* Patient has inadequate venous access for repeated blood draw required for PRP preparation.
* Concurrent participation in a clinical trial in which an investigational agent is used.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Wound Closure | 20 weeks
  The primary objective of this trial is to evaluate increasing the proportion of wounds with complete closure within 20 weeks of initial treatment

CONTACTS AND LOCATIONS:
Overall Officials: Louis Thibodeaux, MD,FACCWS, Principal Investigator — TriHealth Hatton Research Institute | Bethesda North Hospital
Locations (1):
- TriHealth Hatton Research Institute | Bethesda North Hospital, Cincinnati, Ohio, United States